CLINICAL TRIAL: NCT01697267
Title: An International, Open Label, Randomised Controlled Trial Comparing Rituximab With Azathioprine as Maintenance Therapy in Relapsing ANCA-associated Vasculitis
Brief Title: Rituximab Vasculitis Maintenance Study
Acronym: RITAZAREM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Collaborators: Arthritis Research UK (Other); Roche Pharma AG (Industry); Genentech, Inc. (Industry); University of Pennsylvania (Other)
Responsible Party: Principal Investigator, David Jayne, Director, Vasculitis and Lupus Clinic, Cambridge University Hospitals NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RITAZAREM; 2012-001102-14 (EudraCT Number)
Record Dates: First submitted 2012-08-31; First posted 2012-10-02 (Estimated); Results first posted 2022-03-18 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-02

CONDITIONS: Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis; Microscopic Polyangiitis; Wegener Granulomatosis
Keywords: vasculitis; ANCA vasculitis; microscopic polyangiitis; granulomatosis; Wegener's; AAV; vasculitides
MeSH Terms: conditions — Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis; Microscopic Polyangiitis; Granulomatosis with Polyangiitis; Vasculitis | interventions — Rituximab; Azathioprine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rituximab Maintenance (Experimental): Rituximab maintenance: 1g at 4, 8, 12, 16 & 20 months with standardised steroid taper
  Interventions: Biological: Rituximab
- Azathioprine Maintenance (Active Comparator): Azathioprine Maintenance: 2mg/kg/day with standardised steroid taper, from month 4 (randomisation) (200 mg maximum daily dose). Azathioprine withdrawn at month 27.
  Interventions: Drug: Azathioprine

INTERVENTIONS:
Biological: Rituximab — Rituximab IV infusion 1000 mg x 1 dose at months 4, 8, 12, 16 and 20 and glucocorticoids. Four - six hour infusion. Treatment with rituximab will cease at month 20.
  Other Names: Rituxan; MabThera
  Arms: Rituximab Maintenance
Drug: Azathioprine — Oral dosage form. Target dose is 2mg/kg; maximum daily dose is 200mg. This should be continued until month 24. The dose should then by reduced by 50% and azathioprine completely withdrawn at month 27.
  The dose should be rounded down to the nearest 25mg. The dose may vary on alternate days e.g. 100mg one day, 150mg the next for patients on an overall dose of 125mg daily.
  If patients are aged over 60 years, reduce the dose by 25%. If patients are aged over 75 years, reduce the dose by 50%.
  Other Names: Imuran
  Arms: Azathioprine Maintenance

SUMMARY:
Rituximab is now established as an effective drug for anti-neutrophil cytoplasmic antibody (ANCA) vasculitis following major European and US trials reported in 2010. After a time, its effect wears off and the disease can return. This occurs in at least half of patients within 2 years of receiving Rituximab. A preliminary study in Cambridge has suggested that repeating rituximab every six months stops the disease returning and is safe.

The RITAZAREM trial will find out whether repeating rituximab stops vasculitis returning and whether it works better than the older treatments, azathioprine or methotrexate. It will also tell us how long patients remain well after the repeated rituximab treatments are stopped, and if repeated rituximab is safe. We should also learn useful information about the effects of rituximab on quality of life and economic measures. The trial results will help decide the best treatment for future patients who have their vasculitis initially treated with rituximab.

RITAZAREM aims to recruit patients with established ANCA vasculitis whose disease has come back 'relapsing vasculitis'. All patients will be treated with rituximab and steroids and we anticipate that most will respond well. If their disease is under reasonable control after four months, further treatment with either rituximab (a single dose ever four months for two years) or azathioprine tablets will be chosen randomly. The patients in the rituximab and azathioprine groups will then be compared. Patients will be in the trial for four years.

The study has been designed by members of the European Vasculitis Study group (EUVAS) and the Vasculitis Clinical Research Consortium (VCRC). It will include 190 participants from 30 hospitals in Europe, the USA, Australia and Mexico.

RITAZAREM is being funded by Arthritis Research UK, the U.S. National Institutes of Health and by Roche/Genentech.

DETAILED DESCRIPTION:
Patients will be recruited at the time of relapse. All will receive rituximab 375 mg/m2/week x 4 and glucocorticoids.

Those patients that achieve disease control (BVAS/WG ≤ 1 and daily prednisone dose ≤ 10 mg) by month 4 will be randomised to the rituximab or control remission maintenance groups.

Treatment is protocolised for the entire duration of the study, until the common close date, when the final patient recruited has completed 36 months within the study or until the patient has completed 48 months on study whichever the sooner. Patients in the rituximab arm will receive treatment until month 20, and those in the azathioprine arm until month 27.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of AAV [granulomatosis with polyangiitis or microscopic polyangiitis], according to the definitions of the Chapel Hill Consensus Conference
2. Current or historical PR3/MPO ANCA positivity by ELISA
3. Disease relapse defined by one major or three minor disease activity items on the Birmingham Vasculitis Activity Score for Wegeners (BVAS/WG), in patients that have previously achieved remission following at least 3 months of induction therapy, with a combination of glucocorticoids and an immunosuppressive agent (cyclophosphamide or methotrexate or rituximab or mycophenolate mofetil)
4. Written informed consent

Exclusion Criteria:

1. Age < 15 years (age < 18 years at centres that do not treat paediatric patients)
2. Exclusions related to medication:

   Previous therapy with:
   1. Any biological B cell depleting agent (such as rituximab or belimumab) within the past 6 months
   2. Alemtuzumab or anti-thymocyte globulin (ATG) within the last 12 months
   3. IVIg, infliximab, etanercept, adalimumab, abatacept or plasma exchange in past 3 months
   4. Any investigational agent within 28 days of screening, or 5 half lives of the investigational drug (whichever is longer)
3. Exclusions related to general health:

   1. Significant or uncontrolled medical disease not related to AAV, which in the investigators opinion would preclude patient participation
   2. Presence of another multisystem autoimmune disease, including Churg Strauss syndrome, systemic lupus erythematosus, anti-GBM disease, or cryoglobulinaemic vasculitis,
   3. Any concomitant condition anticipated to likely require greater than 4 weeks per year of oral or systemic glucocorticoid use and which would preclude compliance with the glucocorticoid protocol (e.g. poorly-controlled asthma, COPD, psoriasis, or inflammatory bowel disease).
   4. History of severe allergic or anaphylactic reactions to humanised or murine chimeric monoclonal antibodies
   5. Known infection with HIV (HIV testing will not be a requirement for trial entry); a past or current history of hepatitis B virus or hepatitis C virus infection.
   6. Ongoing or recent (last 12 months) evidence of active tuberculosis or known active infection (screening for tuberculosis is part of "standard of care" in patients with established AAV) or evidence of untreated latent tuberculosis. Screening for tuberculosis is as per local practice.
   7. History of malignancy within the past five years or any evidence of persistent malignancy, except fully excised basal cell or squamous cell carcinomas of the skin, or cervical carcinoma in situ which has been treated or excised in a curative procedure.
   8. Pregnancy or inadequate contraception in pre-menopausal women
   9. Breast feeding or lactating
4. Exclusion criteria related to laboratory parameters:

   1. Bone marrow suppression as evidenced by a total white count < 4 x109/l, haemoglobin < 7 gm/dl or platelet count < 100,000/μl
   2. Aspartate aminotransferase or alanine aminotransferase or amylase > 2.5 times the upper limit of normal, unless attributed to vasculitis

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2018-11-22 (Actual); Study Completion 2019-11-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Jayne, Study Chair — Cambridge University Hospitals NHS Foundation Trust; Peter Merkel, Study Chair — University of Pennsylvania
Locations (38):
- United States (9):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Hospital for Special Surgery, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Utah, Salt Lake City, Utah
- Australia (3):
  - Canberra Hospital, Garran, Australian Capital Territory
  - Royal Brisbane & Women's Hospital, Herston, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
- Canada (2):
  - St. Joseph's Healthcare, Hamilton, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
- General Faculty Hospital, Prague, Czechia
- Cork University Hospital, Cork, Ireland
- University Hospital of Parma, Parma, Italy
- Japan (7):
  - Okayama University, Kita-ku, Okayama-ken
  - Chiba University, Chiba
  - Kitano Hospital, Kyoto
  - University of Miyazaki, Miyazaki
  - Teikyo University, Tokyo
  - Tokyo Metropolitan Geriatric, Tokyo
  - Kyorin University school of medicine, Tokyo
- New Zealand (2):
  - Auckland City Hospital, Grafton, Auckland
  - North Shore Hospital, Westlake, Auckland
- Karolinska University Hospital, Stockholm, Sweden
- United Kingdom (11):
  - Leicester General Hospital, Leicester, Leicestershire
  - Queen Elizabeth Hospital, Birmingham
  - Brighton and Sussex University Hospitals, Brighton
  - Addenbrooke's Hospital, Cambridge
  - Russells Hall Hospital, Dudley
  - Ipswich Hospital, Ipswich
  - Chapel Allerton Hospital, Leeds
  - Imperial College, London
  - James Cook University Hospital, Middlesbrough
  - Queen's Medical Centre Campus, Nottingham University Hosp, Nottingham
  - University of Oxford, Oxford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Watts RA, Suppiah R, Merkel PA, Luqmani R. Systemic vasculitis--is it time to reclassify? Rheumatology (Oxford). 2011 Apr;50(4):643-5. doi: 10.1093/rheumatology/keq229. Epub 2010 Jul 20. No abstract available. PMID 20647295
- [Background] Falk RJ, Jennette JC. ANCA disease: where is this field heading? J Am Soc Nephrol. 2010 May;21(5):745-52. doi: 10.1681/ASN.2009121238. Epub 2010 Apr 15. PMID 20395376
- [Background] Watts RA, Scott DG. Epidemiology of the vasculitides. Curr Opin Rheumatol. 2003 Jan;15(1):11-6. doi: 10.1097/00002281-200301000-00003. PMID 12496504
- [Background] Booth AD, Almond MK, Burns A, Ellis P, Gaskin G, Neild GH, Plaisance M, Pusey CD, Jayne DR; Pan-Thames Renal Research Group. Outcome of ANCA-associated renal vasculitis: a 5-year retrospective study. Am J Kidney Dis. 2003 Apr;41(4):776-84. doi: 10.1016/s0272-6386(03)00025-8. PMID 12666064
- [Background] Jayne D, Rasmussen N, Andrassy K, Bacon P, Tervaert JW, Dadoniene J, Ekstrand A, Gaskin G, Gregorini G, de Groot K, Gross W, Hagen EC, Mirapeix E, Pettersson E, Siegert C, Sinico A, Tesar V, Westman K, Pusey C; European Vasculitis Study Group. A randomized trial of maintenance therapy for vasculitis associated with antineutrophil cytoplasmic autoantibodies. N Engl J Med. 2003 Jul 3;349(1):36-44. doi: 10.1056/NEJMoa020286. PMID 12840090
- [Background] de Groot K, Harper L, Jayne DR, Flores Suarez LF, Gregorini G, Gross WL, Luqmani R, Pusey CD, Rasmussen N, Sinico RA, Tesar V, Vanhille P, Westman K, Savage CO; EUVAS (European Vasculitis Study Group). Pulse versus daily oral cyclophosphamide for induction of remission in antineutrophil cytoplasmic antibody-associated vasculitis: a randomized trial. Ann Intern Med. 2009 May 19;150(10):670-80. doi: 10.7326/0003-4819-150-10-200905190-00004. PMID 19451574
- [Background] De Groot K, Rasmussen N, Bacon PA, Tervaert JW, Feighery C, Gregorini G, Gross WL, Luqmani R, Jayne DR. Randomized trial of cyclophosphamide versus methotrexate for induction of remission in early systemic antineutrophil cytoplasmic antibody-associated vasculitis. Arthritis Rheum. 2005 Aug;52(8):2461-9. doi: 10.1002/art.21142. PMID 16052573
- [Background] Wegener's Granulomatosis Etanercept Trial (WGET) Research Group. Etanercept plus standard therapy for Wegener's granulomatosis. N Engl J Med. 2005 Jan 27;352(4):351-61. doi: 10.1056/NEJMoa041884. PMID 15673801
- [Background] Seo P, Min YI, Holbrook JT, Hoffman GS, Merkel PA, Spiera R, Davis JC, Ytterberg SR, St Clair EW, McCune WJ, Specks U, Allen NB, Luqmani RA, Stone JH; WGET Research Group. Damage caused by Wegener's granulomatosis and its treatment: prospective data from the Wegener's Granulomatosis Etanercept Trial (WGET). Arthritis Rheum. 2005 Jul;52(7):2168-78. doi: 10.1002/art.21117. PMID 15986348
- [Background] Reff ME, Carner K, Chambers KS, Chinn PC, Leonard JE, Raab R, Newman RA, Hanna N, Anderson DR. Depletion of B cells in vivo by a chimeric mouse human monoclonal antibody to CD20. Blood. 1994 Jan 15;83(2):435-45. PMID 7506951
- [Background] Jones RB, Tervaert JW, Hauser T, Luqmani R, Morgan MD, Peh CA, Savage CO, Segelmark M, Tesar V, van Paassen P, Walsh D, Walsh M, Westman K, Jayne DR; European Vasculitis Study Group. Rituximab versus cyclophosphamide in ANCA-associated renal vasculitis. N Engl J Med. 2010 Jul 15;363(3):211-20. doi: 10.1056/NEJMoa0909169. PMID 20647198
- [Background] Stone JH, Merkel PA, Spiera R, Seo P, Langford CA, Hoffman GS, Kallenberg CG, St Clair EW, Turkiewicz A, Tchao NK, Webber L, Ding L, Sejismundo LP, Mieras K, Weitzenkamp D, Ikle D, Seyfert-Margolis V, Mueller M, Brunetta P, Allen NB, Fervenza FC, Geetha D, Keogh KA, Kissin EY, Monach PA, Peikert T, Stegeman C, Ytterberg SR, Specks U; RAVE-ITN Research Group. Rituximab versus cyclophosphamide for ANCA-associated vasculitis. N Engl J Med. 2010 Jul 15;363(3):221-32. doi: 10.1056/NEJMoa0909905. PMID 20647199
- [Background] Jones RB, Ferraro AJ, Chaudhry AN, Brogan P, Salama AD, Smith KG, Savage CO, Jayne DR. A multicenter survey of rituximab therapy for refractory antineutrophil cytoplasmic antibody-associated vasculitis. Arthritis Rheum. 2009 Jul;60(7):2156-68. doi: 10.1002/art.24637. PMID 19565480
- [Derived] Smith RM, Jones RB, Specks U, Bond S, Nodale M, Al-Jayyousi R, Andrews J, Bruchfeld A, Camilleri B, Carette S, Cheung CK, Derebail V, Doulton T, Ferraro A, Forbess L, Fujimoto S, Furuta S, Gewurz-Singer O, Harper L, Ito-Ihara T, Khalidi N, Klocke R, Koening C, Komagata Y, Langford C, Lanyon P, Luqmani R, McAlear C, Moreland LW, Mynard K, Nachman P, Pagnoux C, Peh CA, Pusey C, Ranganathan D, Rhee RL, Spiera R, Sreih AG, Tesar V, Walters G, Wroe C, Jayne D, Merkel PA; RITAZAREM co-investigators. Rituximab versus azathioprine for maintenance of remission for patients with ANCA-associated vasculitis and relapsing disease: an international randomised controlled trial. Ann Rheum Dis. 2023 Jul;82(7):937-944. doi: 10.1136/ard-2022-223559. Epub 2023 Mar 23. PMID 36958796
- [Derived] Gopaluni S, Smith RM, Lewin M, McAlear CA, Mynard K, Jones RB, Specks U, Merkel PA, Jayne DR; RITAZAREM Investigators. Rituximab versus azathioprine as therapy for maintenance of remission for anti-neutrophil cytoplasm antibody-associated vasculitis (RITAZAREM): study protocol for a randomized controlled trial. Trials. 2017 Mar 7;18(1):112. doi: 10.1186/s13063-017-1857-z. PMID 28270229

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 188 enrolled participants, 170 met the criteria for randomisation and were randomised for treatment.
Groups:
- Azathioprine Maintenance: Azathioprine Maintenance: 2mg/kg/day with standardised steroid taper, from month 4 (randomisation) (200 mg maximum daily dose). Azathioprine withdrawn at month 27.
  Azathioprine: Oral dosage form. Target dose is 2mg/kg; maximum daily dose is 200mg. This should be continued until month 24. The dose should then by reduced by 50% and azathioprine completely withdrawn at month 27.
  The dose should be rounded down to the nearest 25mg. The dose may vary on alternate days e.g. 100mg one day, 150mg the next for patients on an overall dose of 125mg daily.
  If patients are aged over 60 years, reduce the dose by 25%. If patients are aged over 75 years, reduce the dose by 50%.
Period: Overall Study
Arm/Group | Rituximab Maintenance | Azathioprine Maintenance
Started | 85 | 85
Month 24 | 78 | 78
Completed | 71 | 70
Not Completed | 14 | 15
Not completed — Death | 3 | 1
Not completed — Withdrawal by Subject | 5 | 5
Not completed — Adverse Event | 2 | 1
Not completed — Lost to Follow-up | 2 | 4
Not completed — Physician Decision | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rituximab Maintenance | Azathioprine Maintenance | Total
Number analyzed (Participants) | 85 | 85 | 170
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 54 | 51 | 105
  >=65 years | 31 | 34 | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.1 (15.1) | 58.6 (13.9) | 57.8 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 44 | 86
  Male | 43 | 41 | 84
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 78 | 77 | 155
  Black | 0 | 0 | 0
  Asian | 5 | 5 | 10
  Hispanic | 2 | 1 | 3
  Other | 0 | 2 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 13 | 11 | 24
  Sweden | 3 | 2 | 5
  United States | 26 | 22 | 48
  Czechia | 0 | 1 | 1
  Japan | 2 | 2 | 4
  United Kingdom | 36 | 42 | 78
  Australia | 5 | 5 | 10
ANCA type [Count of Participants; unit: Participants] — Anti-neutrophil cytoplasm antibodies (ANCA) are autoantibodies that target a type of human white blood cell called neutrophils, which are important in health for fighting infection partly through the release of toxic substances that destroy bacteria. In ANCA-associated vasculitis, ANCA specifically bind to two proteins that are normally found in the fluid within the neutrophil (cytoplasm). The two proteins are called proteinase 3 (PR3) and myeloperoxidase (MPO) which can be measured by ELISA (Enzyme-Linked Immunosorbant Assay).
  Participants
    anti-PR3 | 61 | 62 | 123
    anti-MPO | 24 | 23 | 47
Prednisone Induction Regimen [Count of Participants; unit: Participants] — Patients will be stratified at the time of randomisation according to selected prednisone induction regimen: 1A higher dose induction regimen or
  1B lower dose induction regimen to take into consideration variability in disease severity and local GC prescribing.
  Participants
    1A (starting dose 1mg/kg/day) | 24 | 24 | 48
    1B (starting dose 0.5mg/kg/day) | 61 | 61 | 122
Relapse type [Count of Participants; unit: Participants] — Major relapse (severe): The development of a new or recurrent major disease activity item using the BVAS/WG assessment tool Minor relapse (non-severe): Any increase in disease activity that does not meet the definition of Major Relapse
  Participants
    Severe | 52 | 54 | 106
    Non-severe | 33 | 31 | 64

OUTCOME MEASURES:

1. Primary Outcome: Relapse-free Survival
Description: The primary efficacy outcome measure of the trial is relapse-free survival, where a relapse is either major or minor. The primary analysis will be a Cox regression model adjusted for the stratification factors (ANCA type, relapse severity and prednisone induction regimen) for the difference in the distribution of relapse-free survival between the rituximab arm and the azathioprine (control) arm (two-sided at α-level of 5%).
Time Frame: Any patients who have not relapsed at up to a maximum of 4 years will be censored.
Measure: Number; unit: participants
Arm/Group | Rituximab Maintenance | Azathioprine Maintenance
Number analyzed (Participants) | 85 | 85
participants
  Total number of patients with a relapse | 38 | 60
  Total number of patients with a relapse during treatment | 13 | 32
  Total number of patients with a relapse post treatment | 25 | 28

2. Secondary Outcome: Number of Participants in Remission at 24 and 48 Months
Description: Proportion of patients who maintain remission at 24 and 48 months
Time Frame: 24 and 48 months
Measure: Count of Participants; unit: Participants
Arm/Group | Rituximab Maintenance | Azathioprine Maintenance
Number analyzed (Participants) | 85 | 85
Participants
  Month 24 | 73 | 70
  Month 48 | 54 | 44

3. Secondary Outcome: Combined Damage Assessment Score (Disease Related Damage Assessment)
Description: Cumulative accrual of damage as measured by the combined damage assessment score (CDA). Each persistent or new occurrence of damage is given a score of 1. The cumulative accrual of damage is obtained by summing across the different types of damage to get an overall score (max score = 64).
Time Frame: data in Rows represent the change from randomization (month 4) to months 12, 24, 36, and 48.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rituximab Maintenance | Azathioprine Maintenance
Number analyzed (Participants) | 85 | 85
score on a scale
  Randomisation to month 12 | 0.275 (0.656) | 0.337 (0.610)
  Randomisation to month 24 | 0.571 (0.909) | 0.533 (0.777)
  Randomisation to month 36 | 0.676 (0.995) | 0.899 (1.352)
  Randomisation to month 48 | 1.09 (1.18) | 1.38 (1.65)

4. Secondary Outcome: Cumulative GC Exposure
Description: Cumulative glucocorticoid (GC) exposure during the trial. The trial had a common close out date when the final patient reached month 36 in the trial. Patients were followed until month 48 or the common close out date, whichever happened sooner. Therefore, follow up varied between 36 and 48 months. Cumulative glucocorticoid exposure is presented as a dose in mg for during the treatment period (up to month 24) and across the whole trial (until month 48 or common close out when the final patient reached month 36).
Time Frame: Up to 48 months
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Rituximab Maintenance | Azathioprine Maintenance
Number analyzed (Participants) | 85 | 85
mg
  Overall (randomisation to end of trial) | 3717 (3318) | 4780 (3387)
  Maintenance treatment period (randomisation to month 24) | 2184 (1100) | 2426 (1324)

5. Secondary Outcome: Severe Adverse Event Rate
Description: Severe adverse event (SAE) rate
Time Frame: Up to 48 months
Measure: Count of Participants; unit: Participants
Arm/Group | Rituximab Maintenance | Azathioprine Maintenance
Number analyzed (Participants) | 85 | 85
Participants | 37 | 48

6. Secondary Outcome: Infection Rates
Description: Infection (treated with intravenous or oral antibiotics) rates
Time Frame: Up to 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Rituximab Maintenance | Azathioprine Maintenance
Number analyzed (Participants) | 85 | 85
Participants | 54 | 62

7. Secondary Outcome: Health-related Quality of Life Using the SF-36 Physical Composite
Description: The 36-Item Short Form Health Survey (SF-36) is a set of generic, coherent, and easily administered quality-of-life measures. Scores for the scale range from 0-100 and transformed to have a mean of 50 and SD of 10 in the reference population, with higher scores indicating a better Health-related Quality of Life.
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rituximab Maintenance | Azathioprine Maintenance
Number analyzed (Participants) | 83 | 81
score on a scale | 36.7 (15.4) | 36.1 (14.1)

8. Secondary Outcome: Health-related Quality of Life Using the SF-36 Mental Composite
Description: as for outcome 7
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rituximab Maintenance | Azathioprine Maintenance
Number analyzed (Participants) | 83 | 81
score on a scale | 51.8 (11.3) | 51.0 (11.4)

9. Secondary Outcome: Health-related Quality of Life Using the SF-36 Physical Composite
Description: as for outcome 7
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rituximab Maintenance | Azathioprine Maintenance
Number analyzed (Participants) | 80 | 80
score on a scale | 38.2 (15.2) | 34.6 (15.0)

10. Secondary Outcome: Health-related Quality of Life Using the SF-36 Mental Composite
Description: as for outcome 7
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rituximab Maintenance | Azathioprine Maintenance
Number analyzed (Participants) | 80 | 80
score on a scale | 50.8 (12.4) | 51.9 (11.6)

11. Secondary Outcome: Health-related Quality of Life Using the SF-36 Physical Composite
Description: as for outcome 7
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rituximab Maintenance | Azathioprine Maintenance
Number analyzed (Participants) | 77 | 70
score on a scale | 36.7 (15.8) | 35.6 (14.5)

12. Secondary Outcome: Health-related Quality of Life Using the SF-36 Mental Composite
Description: as for outcome 7
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rituximab Maintenance | Azathioprine Maintenance
Number analyzed (Participants) | 77 | 70
score on a scale | 51.9 (11.9) | 53.5 (10.7)

13. Secondary Outcome: Health-related Quality of Life Using the SF-36 Physical Composite
Description: as for outcome 7
Time Frame: 36 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rituximab Maintenance | Azathioprine Maintenance
Number analyzed (Participants) | 74 | 69
score on a scale | 34.6 (15.9) | 33.8 (15.6)

14. Secondary Outcome: Health-related Quality of Life Using the SF-36 Mental Composite
Description: as for outcome 7
Time Frame: 36 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rituximab Maintenance | Azathioprine Maintenance
Number analyzed (Participants) | 74 | 69
score on a scale | 52.3 (12.5) | 51.8 (10.8)

15. Secondary Outcome: Health-related Quality of Life Using the SF-36 Physical Composite
Description: as for outcome 7
Time Frame: 48 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rituximab Maintenance | Azathioprine Maintenance
Number analyzed (Participants) | 55 | 51
score on a scale | 35.8 (14.9) | 35.0 (16.3)

16. Secondary Outcome: Health-related Quality of Life Using the SF-36 Mental Composite
Description: as for outcome 7
Time Frame: 48 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rituximab Maintenance | Azathioprine Maintenance
Number analyzed (Participants) | 55 | 51
score on a scale | 50.9 (13.0) | 53.9 (9.8)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for up to 48 months or until the last patient recruited reached Month 36.
Arm/Group | Rituximab Maintenance | Azathioprine Maintenance
All-Cause Mortality (participants affected / at risk) | 3/85 | 1/85
Serious Adverse Events (participants affected / at risk) | 19/85 | 31/85
Other Adverse Events (participants affected / at risk) | 42/85 | 43/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rituximab Maintenance (N=85) | Azathioprine Maintenance (N=85)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 2 (2) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Periorbital oedema (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Oesophageal spasm (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enterovesical fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Perforated ulcer (General disorders) | 1 (1) | 0 (0)
Stenosis (General disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 2 (2)
Pulmonary vasculitis (Immune system disorders) | 0 (0) | 1 (1)
Vasculitis (Immune system disorders) | 4 (13) | 9 (13)
Appendicitis (Infections and infestations) | 2 (2) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 2 (2)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Dacryocystitis (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 2 (2) | 3 (3)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2)
Peritonitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 5 (5) | 3 (3)
Pneumonia klebsiella (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia viral (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Periorbital abscess (Infections and infestations) | 1 (1) | 0 (0)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1) | 3 (3)
Metapneumovirus infection (Infections and infestations) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1)
Accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Intra-abdominal haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Medical observation (Investigations) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Myasthenia gravis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myasthenia gravis crisis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pubis fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bladder papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Sarcoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Colon neoplasm 1 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Anal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Sleep apnoea syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Subdural haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Conversion disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 4 (4)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Laryngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Aortic valve replacement (Surgical and medical procedures) | 1 (1) | 0 (0)
Bunion operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Cholecystectomy (Surgical and medical procedures) | 1 (1) | 1 (1)
Colostomy closure (Surgical and medical procedures) | 0 (0) | 1 (1)
Dacryocystorhinostomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Hip arthroplasty (Surgical and medical procedures) | 2 (2) | 3 (3)
Knee arthroplasty (Surgical and medical procedures) | 2 (2) | 1 (1)
Lung lobectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Renal transplant (Surgical and medical procedures) | 1 (1) | 0 (0)
Spinal decompression (Surgical and medical procedures) | 0 (0) | 1 (1)
Renal and pancreas transplant (Surgical and medical procedures) | 1 (1) | 0 (0)
Sigmoidectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Cardiac ablation (Surgical and medical procedures) | 0 (0) | 1 (1)
Infusion (Surgical and medical procedures) | 0 (0) | 1 (1)
Colporrhaphy (Surgical and medical procedures) | 1 (1) | 0 (0)
Thyroidectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Joint resurfacing surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
Vascular anastomosis (Surgical and medical procedures) | 0 (0) | 1 (1)
Epistaxis (Vascular disorders) | 0 (0) | 2 (2)
Haemoptysis (Vascular disorders) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Vascular disorders) | 0 (0) | 1 (1)
Vascular injury (Vascular disorders) | 1 (1) | 0 (0)
Vascular pseudoaneurysm (Vascular disorders) | 0 (0) | 1 (1)
Haemorrhage (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rituximab Maintenance (N=85) | Azathioprine Maintenance (N=85)
Malaise (General disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bacterial dacryocystitis (Infections and infestations) | 0 (0) | 1 (1)
Bacterial infection (Infections and infestations) | 2 (2) | 0 (0)
Beta haemolytic streptococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis haemophilus (Infections and infestations) | 2 (2) | 0 (0)
Cellulitis (Infections and infestations) | 3 (3) | 5 (5)
Cellulitis orbital (Infections and infestations) | 0 (0) | 1 (1)
Citrobacter infection (Infections and infestations) | 1 (1) | 1 (1)
Cystitis escherichia (Infections and infestations) | 1 (1) | 2 (2)
Cystitis klebsiella (Infections and infestations) | 0 (0) | 1 (1)
Enterococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 3 (3) | 2 (2)
Haemophilus infection (Infections and infestations) | 2 (2) | 4 (4)
Klebsiella infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia haemophilus (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia klebsiella (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia pneumococca (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia pseudomonal (Infections and infestations) | 1 (1) | 0 (0)
Proteus infection (Infections and infestations) | 1 (1) | 0 (0)
Pseudomonas bronchitis (Infections and infestations) | 2 (2) | 1 (1)
Pseudomonas infection (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal impetigo (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 3 (3) | 2 (2)
Tonsillitis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection enterococcal (Infections and infestations) | 2 (2) | 1 (1)
Body tinea (Infections and infestations) | 1 (1) | 0 (0)
Candida infection (Infections and infestations) | 1 (1) | 1 (1)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 2 (2) | 1 (1)
Tinea infection (Infections and infestations) | 1 (1) | 0 (0)
Tinea pedis (Infections and infestations) | 0 (0) | 1 (1)
Vulvovaginal candidiasis (Infections and infestations) | 1 (1) | 2 (2)
Vulvovaginal mycotic infection (Infections and infestations) | 2 (2) | 0 (0)
Bronchitis (Infections and infestations) | 2 (2) | 0 (0)
Conjunctivitis (Infections and infestations) | 2 (2) | 2 (2)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 5 (5) | 4 (4)
Eye infection (Infections and infestations) | 0 (0) | 2 (2)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 2 (2)
Lower respiratory tract infection (Infections and infestations) | 2 (2) | 7 (7)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Mastoiditis (Infections and infestations) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 2 (2) | 0 (0)
Pharyngitis (Infections and infestations) | 2 (2) | 2 (2)
Pneumonia (Infections and infestations) | 3 (3) | 1 (1)
Prostate infection (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 19 (19) | 31 (31)
Root canal infection (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 15 (15) | 10 (10)
Skin infection (Infections and infestations) | 5 (5) | 4 (4)
Systemic infection (Infections and infestations) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 1 (1) | 2 (2)
Tooth infection (Infections and infestations) | 3 (3) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 17 (17) | 17 (17)
Urinary tract infection (Infections and infestations) | 9 (9) | 7 (7)
Herpes simplex (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 1 (1)
Oral herpes (Infections and infestations) | 0 (0) | 2 (2)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0)
Varicella zoster virus infection (Infections and infestations) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Streptococcus test positive (Investigations) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rosacea (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-07-12): https://cdn.clinicaltrials.gov/large-docs/67/NCT01697267/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-25): https://cdn.clinicaltrials.gov/large-docs/67/NCT01697267/SAP_001.pdf